CLINICAL TRIAL: NCT04829071
Title: Cognition as a Moderator of Motor Learning Post-stroke
Brief Title: Cognition and Motor Learning Post-stroke
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kristan Leech, Principal Investigator, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APP-21-00898
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Stroke; CVA (Cerebrovascular Accident)
Keywords: stroke; walking; rehabilitation; cognition
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluating motor learning and brain structures post-stroke (Experimental): We will use a single arm design to determine the impact of post-stroke cognitive impairment on two forms of motor learning (implicit and explicit) and evaluate the structural integrity of relevant brain structures in 65 individuals post stroke
  Interventions: Behavioral: Explicit motor learning; Behavioral: Implicit motor learning

INTERVENTIONS:
Behavioral: Explicit motor learning — Participants will be provided with visual feedback of their right and left step lengths on a screen in front of a treadmill.
Behavioral: Implicit motor learning — Participants will walk on a treadmill that drives their right and left legs to move at two different speeds.

SUMMARY:
This project seeks to determine how post-stroke cognitive impairment moderates motor learning during walking in older adults with chronic stroke and identify brain structural markers that mediate this relationship. The chosen experimental design integrates biomechanical analyses, neuropsychological assessments, and brain imaging techniques to determine the impact of post-stroke cognitive impairment severity on two forms of motor learning (explicit and implicit) and examine the role of the dorsolateral prefrontal cortex in the relationship between cognition and explicit motor learning. Ultimately, this work may lead to the development of a more comprehensive, effective treatment approach to improve walking dysfunction in older adults post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke
* Stroke occurred more than 6 months prior
* Paresis confined to one side
* Independently ambulatory (including the use of assistive devices)
* Able to walk for 5 minutes without stopping
* Answers no to all general health questions on the PAR-Q+
* Willingness to complete study procedures

Exclusion Criteria:

* Brainstem or cerebellar stroke
* Aphasia (expressive, receptive, or global)
* Any major musculoskeletal or non-stroke neurological condition that interferes with the assessment of sensorimotor or cognitive function
* Metal in the head (except in the mouth), implanted cranial or thoracic devices that violate MRI safety regulations
* Uncontrolled hypertension (>160/110mmHg)
* Concurrent physical therapy
* Claustrophobia
* Significant cognitive deficit or dementia (<20 on MoCA)
* Inability to give informed consent

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2026-08-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
step length asymmetry - change in performance | Measured at three timepoints of interest within each testing session: baseline and at the beginning and end of the interventions; participants will complete 2 testing sessions over approximately 1 months
  characterized as a comparison between the right and left step lengths; captured to quantify change in performance with biofeedback or split belt walking

SECONDARY OUTCOMES:
step length asymmetry - immediate retention | Measured after motor learning in each testing session; participants will complete 2 testing sessions over approximately 1 months
  characterized as a comparison between the right and left step lengths; captured to quantify the retention of a newly learned walking pattern

CONTACTS AND LOCATIONS:
Overall Officials: Kristan Leech, PT, DPT, PhD, Principal Investigator — University of Southern California
Locations (1):
- Center for Health Professions, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data from our research that underlie results in a publication will be made available on the Open Science Framework.
Supporting Information: Analytic Code
Time Frame: data will be made available 6 months after publication